CLINICAL TRIAL: NCT02778854
Title: Liquid Biopsy for Detection of Driver Mutation in Diagnostic and Prognostic of NSCLC
Brief Title: Liquid Biopsy for Detection of Driver Mutation in NSCLC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Chen Liang_An, MD,PHD, Chinese PLA General Hospital
Other Study IDs: S2015-099-01
Record Dates: First submitted 2016-05-10; First posted 2016-05-20 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC; liquid biopsy; driver mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — body fluid
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- cohort 1: Participants are recruited for diagnostic test
  Interventions: Genetic: detection of driver mutation
- cohort 2: participants are recruited for follow-up
  Interventions: Genetic: detection of driver mutation

INTERVENTIONS:
Genetic: detection of driver mutation — participants are received gene detection via the liquid biopsy

SUMMARY:
The purpose of this study is to evaluate the diagnostic and prognostic efficacy of liquid biopsy in different specimens and in different methods compared with tissue detection .

DETAILED DESCRIPTION:
Collect plasma and other specimens from patients who are newly diagnosed with NSCLC or with drug-resistant and plan to receive gene detection to complete the diagnostic test for liquid biopsy .Participants who come from diagnostic test and plan to receive tyrosine kinase inhibitors (TKI) therapy will be collected plasma and other specimens every month during the regiments and monitor the changes of driver motion to predict the prognosis of targeted therapy.

ELIGIBILITY:
cohort 1

Inclusion Criteria:

* patients newly diagnosed with NSCLC confirmed by tissue biopsy and going to receive the detection of gene mutation or patients have obtained drug-resistance after receiving molecular target therapy and plan to re-biopsy.
* Age ≥ 18 years
* newly diagnosed patients have not received TKI and chemotherapy
* patients who are drug-resistant have not received next-generation TKI

Exclusion Criteria:

* patients who have more than one type of carcinoma
* patients who reject to sign the informed consent from

cohort 2

Inclusion Criteria:

* patients from cohort1 with sensitive driver mutation and plan to receive TKI therapy
* patients will have regular follow-up in Chinese people liberation army general hospital every month.

Exclusion Criteria:

* patients who are refused to provide the informed consent from

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who have been diagnosed with NSCLC and received detection of driver mutation in Chinese PLA general hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-10; Primary Completion 2018-12 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
concordance between tissue and plasma using detection method such as droplet digital PCR(ddPCR) or next generation sequencing(NGS) to detect the driver mutation in NSCLC | 6 months

SECONDARY OUTCOMES:
concordance between tissue and other specimens using detection method such as droplet digital PCR(ddPCR) or next generation sequencing(NGS) to detect the driver mutation in NSCLC | 6 months
changes of driver mutation in quality and quantity in the process of targeted treatment to predict the prognosis | 5 years
Progress-free survival(PFS) in patients who have had driver mutation and received the molecular target therapy | 3 years
  compare the PFS between each participants via the change of driver mutation
Overall survival(OS) in patients who had driver mutation and received the molecular target therapy | 5 years
  compare the OS between each participants via the change of driver mutation

CONTACTS AND LOCATIONS:
Overall Officials: Liang-an Chen, MD,PHD, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- department of respiratory department ,Chinese PLA general hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
considering of personal privacy, the research-related individual participant data do not intend for public sharing.

REFERENCES:
- [Derived] Wu Z, Yang Z, Li CS, Zhao W, Liang ZX, Dai Y, Zhu Q, Miao KL, Cui DH, Chen LA. Differences in the genomic profiles of cell-free DNA between plasma, sputum, urine, and tumor tissue in advanced NSCLC. Cancer Med. 2019 Mar;8(3):910-919. doi: 10.1002/cam4.1935. Epub 2019 Feb 14. PMID 30767431